CLINICAL TRIAL: NCT02155478
Title: Comparison of the Capsular Stability With Two Different IOL Models in Patients With Pseudoexfoliation Syndrome: an Exploratory Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PXF
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMO ZCB00 (Other): AMO ZCB00 IOL (Abbott Medical Optics, United States): a standard IOL
  Interventions: Device: AMO ZCB00 IOL (Abbott Medical Optics, United States): a standard IOL
- ISERT 250 (Active Comparator): ISERT 250 (HOYA, Japan): a standard IOL
  Interventions: Device: ISERT 250 (HOYA, Japan): a standard IOL

INTERVENTIONS:
Device: ISERT 250 (HOYA, Japan): a standard IOL
  Arms: ISERT 250
Device: AMO ZCB00 IOL (Abbott Medical Optics, United States): a standard IOL
  Arms: AMO ZCB00

SUMMARY:
The pseudoexfoliation (PXF syndrome) is caused by production and deposition of extracellular material in the anterior chamber of the eye as well as in other tissues of the body. Approx. 70 million worldwide have a PXF syndrome.

After cataract surgery a decentration and subluxation of the intraocular lens (IOL) happens more frequently than in the general population due to a higher incidence of zonular weakness and an increased capsular fibrotic reaction.

Decentration, tilt and / or rotation of the lens can reduce the quality of vision.

It is believed that the design of the implanted IOL, more precisely the front surface of the IOL has an influence on the extent of capsular fibrosis and contraction. Especially in presence of capsular instability, as it is in patients with Pseudoexfoliation syndrome the design of the IOL has an effect on the post-operative stability.

In this study, two different IOL models are compared in terms of their stability. The "Tecnis 1-piece ZCB00" (AMO, USA), with a concave lowering comprising the lens edge and the "Acrysof SA60AT" (Alcon, USA), with a biconvex design are compared. Forty eyes of 20 patients are planned to be included in this study. One eye receives the "Tecnis ZCB00 1-piece "(AMO, USA), while the other eye receives the"Acrysof SA60AT "(Alcon, USA).

In which eye which IOL is implanted, is assigned by randomization. To measure the decentration, tilt and rotation of the IOL an examination will be performed before the operation and there will be follow-ups one hour after the operation of the first eye, one hour after the operation of the second eye, three months and twelve months after the operation on the second eye. All measurements will be done without touching the eye.

DETAILED DESCRIPTION:
Pseudoexfoliation (PXF) is an age-related disease characterized by production of extracellular material in the anterior segment of the eye and other tissues of the body. While only 0.6% of people between 52 and 65 years are affected, 5% of people between 75 years and 85 years have Pseudoexfoliation syndrome. An estimated 70 million people may have PXF worldwide. PXF can be associated with glaucoma, cataract, reduced pupil dilatation, zonule weakness, and postoperative complications. After cataract surgery decentration and subluxation of the intra-ocular lens (IOL) is more likely in patients with Pseudoexfoliation syndrome due to the higher incidence of zonular weakness as well as the increased capsule fibrotic reaction. It has to be taken into account that an anterior chamber depth (ACD) shift, decentration, tilt or rotation of an IOL could result in a severe reduction in visual quality. For an aspherical IOL, for instance, it is essential not to be decentered and tilted more than 0.4 mm (0.8 mm 7) and 7° (10° 7), respectively. Otherwise it will be outperformed by a spherical IOL. We assume that the design of the IOL, more precisely the design of the anterior surface of the IOL, can influence the degree of capsule fibrosis and contraction, especially in patients who tend to have capsular instability like patients with PXF syndrome. The Tecnis 1-piece ZCB00 (AMO, California, USA), a single-piece hydrophobic acrylic open-loop IOL has its convex anterior surface not up to the edge of the IOL optic, but instead has a concave depression before reaching the edge. Due to this particular shape of the anterior surface, the anterior lens capsule typically only has contact at the IOL optic edge with the remaining central part up to the rhexis edge 'floating' over the optic without contact. Due to this situation, we expect less fibrotic reaction of the capsule because of a lack of contact between the lens epithelial cells of the anterior capsule not transdifferentiating into myofibroblasts and not laying down collagen that result in the typical contraction and whitening of the anterior capsule. On the contrary, another IOL, the ISERT 250 (HOYA, Japan), also a hydrophobic acrylic open-loop IOL, has an anterior surface which is convex all the way to the optic edge resulting in complete contact of the rhexis edge and overlying the anterior capsule on the IOL optic. This may aggravate the anterior lens capsule reaction to the IOL material which may result in more capsular contraction due to pronounced fibrosis of the capsule and in turn results in decentration and or tilt of the IOL.

Aim of this study is to assess the differences of IOL tilt and decentration in patients with pseudoexfoliation syndrome (PXF) with two different IOLs, the Tecnis 1-piece ZCB00, (AMO, USA) and the ISERT 250 (HOYA, Japan), measured with an AS-OCT, Scheimpflug imaging and Purkinjemeter.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* Pseudoexfoliation syndrome
* written informed consent prior to surgery

Exclusion Criteria:

* Relevant ophthalmic diseases that could affect corneal transparency or the ability for fixation of LEDs
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Difference between the two IOLS in postoperative IOL tilt (degrees) and decentration (mm) measured with the Purkinjemeter | 12 months

SECONDARY OUTCOMES:
Horizontal and vertical IOL tilt (in °) evaluated from AS-OCT and Scheimpflug images | 12 months
Change in rhexis diameter (mm in retroillumination foto) | 12 months
Change in anterior chamber depth (in mm) measured with the AC Master | 12 months
Subjective evaluation of IOL - anterior capsule interconnection ( capsule overlapping the IOL optic edge in slitlamp examination) | 12 months
Change in aqueous flare measured with laser flare meter | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Principal Investigator — ViROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital Vienna, Vienna, Austria 1140
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Vienna, Austria